CLINICAL TRIAL: NCT04552106
Title: An Open-label, Single-center, Randomized, Exploratory, Dose-finding Study to Evaluate Short Term Treatment With Different Doses of Oral Powdered Kudzu Root Extract in Women With at Least Mild Menopause Symptoms
Brief Title: Dose Finding Evaluation of Kudzu Root Extract in Women With Menopause Symptoms
Acronym: KUDZU-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol_V1.2_KUDZU
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Menopause

STUDY DESIGN:
Intervention Model Description: Unblinded, single-center, randomized, exploratory, dose-finding study. 1:1:1:1:1 randomisation to 5 groups of different doses for 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Active Comparator): 10 subjects
  Interventions: Dietary Supplement: 3 caps x3/day
- Group 2 (Active Comparator): 10 subjects
  Interventions: Dietary Supplement: 3 caps x2/day
- Group 3 (Active Comparator): 10 subjects
  Interventions: Dietary Supplement: 2 caps x3/day
- Group 4 (Active Comparator): 10 subjects
  Interventions: Dietary Supplement: 2 caps x2/day
- Group 5 (Active Comparator): 10 subjects
  Interventions: Dietary Supplement: 3 caps x1/day

INTERVENTIONS:
Dietary Supplement: 3 caps x3/day — 3 capsules 3 times daily for 28 days
  Arms: Group 1
Dietary Supplement: 3 caps x2/day — 3 capsules 2 times daily for 28 days
  Arms: Group 2
Dietary Supplement: 2 caps x3/day — 2 capsules 3 times daily for 28 days
  Arms: Group 3
Dietary Supplement: 2 caps x2/day — 2 capsules 2 times daily for 28 days
  Arms: Group 4
Dietary Supplement: 3 caps x1/day — 3 capsules 1 times daily for 28 days
  Arms: Group 5

SUMMARY:
The aim of the study is to investigate effects of daily intake of Nordic Kudzu for 28 days in 5 groups of 10 menopausal women with symptoms. Groups:1) 3 capsules x3/day, 2) 3 capsules x2/day, 3) 2 capsules x3/day, 4) 2 capsules x2/day, 5) 3 capsules x1/day. Each capsule equal 1.26 g kudzu root extract. Outcome measures: Serum and urine levels of biochemical marker of bone-degradation, CTX-I, and symptoms of menopause using the Meopause Rating Scale (MRS).

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated informed consent
2. Women in the age between 45 and 60 years considered late peri- (defined as having had a menstrual period more than 3 months ago but less than 12 months ago) or postmenopausal (defined as at least 12 consecutive months without any menstrual flow) at the time of screening
3. Menopause symptoms, defined as a score of at least 5 in the Menopausal Rating Scale (MRS) at screening
4. Body Mass Index between 18 and 40 kg/m2 at the time of screening

Exclusion criteria:

1. Allergy/hypersensitivity/intolerance to any components in the Kudzu herbal extract powder capsules
2. Past or present significant co-morbidity including, but not limited to: Uncontrolled, severe renal, hepatic, cardiovascular, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease
3. History of breast cancer or other malignancy, except adequately treated basal cell or squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ
4. Known history of clinically significant thromboembolism
5. Current alcohol abuse
6. Pregnancy, determined by positive serum human chorionic gonadotropin (hCG) test prior to randomization, except for women considered postmenopausal
7. Breastfeeding women
8. Participation in a study trial with any investigational new drug or food supplement within 3 months prior to the start of the study
9. Clinically significant ECG abnormalities, as judged by the investigator
10. Clinically significant biochemistry abnormalities including but not limited to ALT or AST >2.5 x ULN or other clinically significant liver function parameters, as judged by the investigator
11. Investigator considering the subject inappropriate for inclusion in the study based on medical interview and/or physical examination
12. Use of local or systemic conventional hormone therapy regardless of indication or alternative medication including dietary supplements for the treatment of menopausal symptoms within 28 days prior to randomization.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | 28 days
  Questionaire. 11 likert scales 0-4. Total score ranges: 0-44 (0 indicating no symptoms, 44 indicating max symptoms.
Serum CTX-I | 28 days
  Blood based biomarker of bone resorption
Urine CTX-I | 28 days
  Urine based biomarker of bone resorption

CONTACTS AND LOCATIONS:
Overall Officials: Henning B Nielsen, DMSci, Principal Investigator — Sanos Clinic
Locations (1):
- Sanos Clinic, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No